CLINICAL TRIAL: NCT02868775
Title: A Pilot Study to Determine the Role of Toll-like Receptor-4 Expression in Patients With Interstitial Cystitis/Bladder Pain Syndrome
Brief Title: A Study to Determine the Role of Toll-like Receptor-4 Expression in Patients With Interstitial Cystitis/Bladder Pain Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Philadelphia Urosurgical Associates (Other)
Collaborators: Drexel University College of Medicine (Other)
Responsible Party: Principal Investigator, Kristene Whitmore, Division Head of Female Pelvic Medicine and Reconstructive Surgery, Philadelphia Urosurgical Associates
Other Study IDs: TLR4001
Record Dates: First submitted 2016-08-09; First posted 2016-08-16 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Cystitis, Interstitial; Painful Bladder Syndrome
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Cystoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bladder biopsies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Interstitial cystitis/bladder pain syndrome: These are the patients that will be evaluated in this study.
  Interventions: Procedure: cystoscopy, bladder hydrodistention and bladder biopsy

INTERVENTIONS:
Procedure: cystoscopy, bladder hydrodistention and bladder biopsy

SUMMARY:
This is a prospective pilot study, with a recruitment goal of 60 patients. Patients who are female, above the age of 18, and with a diagnosis of IC/BPS based on clinical criteria and O'Leary Sant ICPI and ICSI scores undergoing cystoscopy, hydrodistention and bladder biopsy will be included. The bladder biopsies will be evaluated for TLR4 expression, and sent for histological assessment of mast cell count. Additionally, data will be collected at baseline, day of surgery, day 7, day 14 and day 28. Data will include validated questionnaires, lower urinary tract symptoms, and recorded pain medication use.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be a candidate for cystoscopy, hydrodistention and bladder biopsy.
2. Participant must have subjective complaints of

   1. urinary urgency, relieved with voiding, OR
   2. urinary frequency; ≥ 8 voids per day, OR
   3. pelvic pain, pressure, or discomfort

2. Gender of subjects: Subjects in this study will be female. Pregnant women and breastfeeding women will be excluded due to unknown risk of study medication on pregnancy and fetus or nursing infants.

3. Age of subjects: Age of subjects will range from 18 to 90 years.

4. Racial and ethnic origin: There are no enrollment restrictions based upon race or ethnic origin. The racial and ethnic distribution of subjects is entirely based on the population of patients at the study site.

5. Other inclusion criteria:

1. Participant must give written informed consent to participate in the study
2. Participant must be able to make decisions for herself
3. Participant must not have had a UTI within 7 days prior to start of the study
4. Female participants who are with a positive pregnancy test

Exclusion Criteria:

To participate in the study subjects must not meet any of the following criteria:

1. Participant is currently pregnant or breastfeeding
2. Participant has a positive urinary pregnancy test at the time of screening
3. Participant is currently or has been on antibiotic therapy with the last 7 days prior to the start of the study
4. Participant is currently in another trial
5. Participant has an active S3 nerve stimulator implanted or has PTNS
6. Participant has had intravesical botulinum toxin injection in 6 months prior to starting the study
7. Participant has grade III or IV pelvic organ prolapse
8. Participant has history of bladder cancer
9. Participant has a neurological disease including, but not limited to, multiple sclerosis, Parkinson's disease, Alzheimer's disease, spinal cord injury, brain injury, stroke or dementia
10. Participant has urinary frequency of less than 8 times/day
11. Participant has bladder or lower ureteral calculi
12. Participant has active genital herpes
13. Participant has urethral diverticulum
14. Participant has chemical cystitis
15. Participant has radiation or tuberculosis cystitis

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients diagnosed with IC/BPS with a minimum O'Leary-Sant score of 8 on the ICSI, as well as 8 on the ICPI who are undergoing cystoscopy, hydrodistention and bladder biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-06 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Toll-like Receptor 4 protein analysis | 1 year
  Determine Toll-like Receptor 4 protein expression with western blot
Toll-like Receptor 4 mRNA expression in bladder biopsy | 1 year
  Determine Toll-like Receptor 4 mRNA expression with quantitative polymerase chain reaction
Toll-like Receptor 4 distribution and localization evaluation | 1 year
  Determine Toll-like Receptor 4 distribution and localization with immunohistochemistry

SECONDARY OUTCOMES:
Bladder symptom evaluation | 28 days
  Utilize O'Leary Sant Interstitial Cystitis Symptom and Problem Indices to evaluate subjective bladder symptom changes
Vaginal symptoms evaluation | 28 days
  Utilize pelvic floor impact questionnaire-7 to evaluate vaginal and pelvic symptoms
Female sexual function | 28 days
  Use female sexual function index questionnaire to evaluate female sexual function
Interstitial cystitis Flares | 28 days
  Patients will record bladder pain scores and changes in urinary urgency with the bladder diary to evaluate flares following cystoscopy, hydrodistention
Patient satisfaction | 28 days
  Use Global response assessment questionnaire
Bladder symptom evaluation | 28 days
  Utilize questionnaire: pelvic floor impact questionnaire-7

CONTACTS AND LOCATIONS:
Locations (1):
- Hahnemann Urogynecology, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No